CLINICAL TRIAL: NCT06348394
Title: Intracardiac Versus Transesophageal Echocardiographic Guidance for Left Atrial Appendage Occlusion
Acronym: ICETEE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 023-318
Record Dates: First submitted 2024-03-12; First posted 2024-04-04 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Left Atrial Appendage Closure

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, parallel controlled, open-label, single center study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intracardiac echocardiography Left atrial appendage closure. (Active Comparator): Intra cardiac echocardiography will be performed prior to left atrial appendage closure.
  Interventions: Other: Intracardiac Echocardiography
- Traditional transesophageal echocardiography guided Left atrial appendage closure (Placebo Comparator): Transesophageal Echocardiography will be performed under general anesthesia.
  Interventions: Other: Intracardiac Echocardiography

INTERVENTIONS:
Other: Intracardiac Echocardiography — Transesophageal echocardiography will be performed under general anesthesia.
  Other Names: Transesophageal Echocardiography

SUMMARY:
This single-center, prospective, randomized study will evaluate the safety and feasibility of Intracardiac echocardiography (ICE)-guided Left atrial appendage closure (LAAC) when compared to the traditional Transesophageal echocardiography (TEE) approach.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the efficacy and safety of using Intracardiac echocardiography (ICE) to guide implantation of percutaneous left atrial appendage closure (LAAC) devices.

Primary endpoints include procedural success following implantation of the left atrial appendage occlusion (LAAO) device. Procedural success specifies that the device should be implanted in the correct position without device related complications and no peri-device leaks >5 mm on color doppler.

Secondary end points include periprocedural complications (such as pericardial effusion/tamponade, stroke, death, vascular complications, and device embolization), procedural characteristics (total duration, fluoroscopy time, contrast volume, Length of hospital stay), cost of hospitalization, in-hospital patient satisfaction, and clinical alterations at 45-day follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed for non-valvular atrial fibrillation with documented paroxysmal, persistent, or permanent NVAF.
2. Deemed to be at high risk of stroke or systemic embolism (SE) defined as a CHADS2 score ≥2 or a CHA2DS2-VASc score ≥3.
3. Patient suitable for OAC with warfarin or DOAC and have appropriate rationale to seek a nonpharmacologic alternative to long-term OAC, meeting commercial LAAO criteria indications.
4. Can undergo appropriate pre-procedural imaging with Computed tomography (CT) or transesophageal echocardiography (TEE).
5. Patient should be able to comply with the protocol.
6. Provide written informed consent before study participation.
7. Ages 18 and above

Exclusion Criteria

1) A patient will be ineligible for inclusion in this study if he or she meets any of the following criteria:

1. Presence of an intracardiac thrombus on the preprocedural TEE or CT.
2. History of previously implanted device for atrial septal defect or patent foramen ovale.
3. Severe LV dysfunction (LVEF < 40%) or greater than moderate valvular heart disease.
4. Enrollment in another study that competes or interferes with this study. Approval to dual enroll must be approved by the other study.
5. Poor clinical condition like cardiogenic shock, which prohibits pre- and post-procedural function tests.
6. Subject with planned cardiac intervention between the time of consenting and up to 60 days post-LAAO.
7. Any other condition or co-morbidity which, in the opinion of the investigator or operator, may pose a significant hazard to the subject if he or she is enrolled in the study.
8. For women of childbearing potential: Pregnant or breastfeeding women or planning pregnancy during the course of the investigation are excluded due to the risks involved in the procedure
9. Children below 18 years, prisoners and patients who are unable to provide consent are excluded.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 444 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2026-12-14 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Procedural success following implantation of the left atrial appendage occlusion (LAAO) device. | Intra op
  Procedural success specifies that the device should be implanted in the correct position measured as:
  Peri-device leaks greater than 5 milliliters on color doppler (Yes/No)

SECONDARY OUTCOMES:
Periprocedural complications | 45 days after the procedure
  Pericardial effusion/tamponade measured as (Yes/No)
Procedural characteristics | 45 days after the procedure
  Total duration measured as number of minutes.
Patient satisfaction | 45 days after the procedure
  Patient satisfaction will be assessed in-hospital by a questionnaire addressing anesthesia-related discomfort.
Periprocedural complications | 45 days after the procedure
  Stroke measured as (Yes/No)
Periprocedural complications | 45 days after the procedure
  Death measured as (Yes/No)
Procedural characteristics | 45 days after the procedure
  Fluoroscopy time measured as number of minutes.
Procedural characteristics | 45 days after the procedure
  Contrast volume measured in milli liters.
Procedural characteristics | 45 days after the procedure
  Length of hospital stay measured as number of days.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor Scott and White Heart Hospital, Plano, Texas, United States

REFERENCES:
- [Background] Reddy VY, Sievert H, Halperin J, Doshi SK, Buchbinder M, Neuzil P, Huber K, Whisenant B, Kar S, Swarup V, Gordon N, Holmes D; PROTECT AF Steering Committee and Investigators. Percutaneous left atrial appendage closure vs warfarin for atrial fibrillation: a randomized clinical trial. JAMA. 2014 Nov 19;312(19):1988-98. doi: 10.1001/jama.2014.15192. PMID 25399274
- [Background] Hemam ME, Kuroki K, Schurmann PA, Dave AS, Rodriguez DA, Saenz LC, Reddy VY, Valderrabano M. Left atrial appendage closure with the Watchman device using intracardiac vs transesophageal echocardiography: Procedural and cost considerations. Heart Rhythm. 2019 Mar;16(3):334-342. doi: 10.1016/j.hrthm.2018.12.013. PMID 30827462
- [Background] Tzikas A, Holmes DR Jr, Gafoor S, Ruiz CE, Blomstrom-Lundqvist C, Diener HC, Cappato R, Kar S, Lee RJ, Byrne RA, Ibrahim R, Lakkireddy D, Soliman OI, Nabauer M, Schneider S, Brachmann J, Saver JL, Tiemann K, Sievert H, Camm AJ, Lewalter T. Percutaneous left atrial appendage occlusion: the Munich consensus document on definitions, endpoints, and data collection requirements for clinical studies. Europace. 2017 Jan;19(1):4-15. doi: 10.1093/europace/euw141. Epub 2016 Aug 18. PMID 27540038